CLINICAL TRIAL: NCT07278128
Title: Evaluation of the Therapeutic Effects of Curcumin on Changes in Lipid, Metabolic, and Hormonal Profiles, Liver Enzyme Activity, and Ultrasonography Morphology of the Liver in Women With Polycystic Ovary Syndrome and Nonalcoholic Fatty Liver Disease: A Double-blind, Placebo-controlled Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fateme Moshirenia (Other)
Responsible Party: Sponsor-Investigator, Fateme Moshirenia, Associate Professor of Reproductive Health and Principal Investigator, Tarbiat Modarres University
Organization: Tarbiat Modarres University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TarbiatModaresU
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Ovary Syndrome (PCOS) With Concurrent Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): curcumin capsules
  Interventions: Drug: Patients (women of reproductive age suffering from non-alcoholic fatty liver with polycystic ovary syndrome) receiving 500 mg curcumin capsules (prepared from the extraction of turmeric in the laborat
- control group (Placebo Comparator): receiving placebo
  Interventions: Drug: Patients (women of reproductive age suffering from non-alcoholic fatty liver with polycystic ovary syndrome) receiving 500 mg curcumin capsules (prepared from the extraction of turmeric in the laborat

INTERVENTIONS:
Drug: Patients (women of reproductive age suffering from non-alcoholic fatty liver with polycystic ovary syndrome) receiving 500 mg curcumin capsules (prepared from the extraction of turmeric in the laborat — Patients (women of reproductive age suffering from non-alcoholic fatty liver with polycystic ovary syndrome) receiving 500 mg curcumin capsules (prepared from the extraction of turmeric in the laboratory of Shahid Beheshti Faculty of Pharmacy in Tehran), twice a day (one gram per day) for three months

SUMMARY:
Background and Objectives:

Polycystic ovary syndrome (PCOS) and nonalcoholic fatty liver disease (NAFLD) commonly co-occur and are associated with insulin resistance, chronic inflammation, and metabolic and hormonal imbalances. Standard drug therapies can cause side effects, so safer and more effective alternatives are needed. This study evaluated whether daily curcumin supplementation could improve lipid, metabolic, hormonal, and liver-related parameters in women of reproductive age with both PCOS and NAFLD.

Study Design and Participants:

This was a double-blind, randomized, placebo-controlled clinical trial conducted at Arash General Women's Hospital. Ninety-four women of reproductive age diagnosed with PCOS and NAFLD were enrolled and randomly assigned to receive curcumin or placebo.

Intervention:

Participants in the intervention group received 1000 mg curcumin daily; the control group received 1000 mg placebo daily. The treatment period was 12 weeks. Measurements were taken at baseline and after 12 weeks.

Key measurements:

Anthropometric measurements, lipid profile (total cholesterol, LDL, HDL, triglycerides), fasting blood glucose, HbA1c, serum testosterone, anti-mullerian hormone (AMH), liver enzymes (AST, ALT, ALP), and liver ultrasound for degree of steatosis.

ELIGIBILITY:
Inclusion criteria:

Women of reproductive age from 18 to 45 years old Women with polycystic ovary syndrome and non-alcoholic fatty liver disease Having two of the three Rotterdam criteria including: Having an ultrasound appearance of polycystic ovaries, having serum hyperandrogenism with/without clinical symptoms related to hyperandrogenism such as acne, hirsutism, acanthosis nigricans, etc., having an ovulation disorder and irregular menstrual cycle. Ability to speak and write in Persian

Exclusion criteria:

-Pregnancy Breastfeeding Using hormonal methods for contraception Having any other diagnosed disease Sensitivity to turmeric History of advanced chronic liver disease Smoking and alcohol use Drug addiction Adrenal hyperplasia that has symptoms similar to polycystic ovary syndrome Kidney failure or any active digestive disorder Other chronic non-metabolic diseases Thyroid disease Hyperprolactinemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-06-22 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Liver ultrasound view (gradient change) | Before the intervention and 48 hours after the end of the intervention
  There is no need to fast, and as soon as possible, the patient is referred to an ultrasound specialist for diagnostic and examination procedures according to specific criteria for examining fatty liver.
Body mass index (BMI) | Before the intervention and 48 hours after the end of the intervention
  Measuring height with a centimeter tape and measuring weight with a digital scale and then entering the obtained values into the formula of weight in kilograms divided by the square of height in meters to calculate the body mass index.
The level of low-density lipoprotein (LDL) | before the intervention and 48 hours after the intervention
  laboratory test
The level of high-density lipoprotein (HDL) | before the intervention and 48 hours after the intervention
  laboratory test
The level of triglyceride (TG) | before the intervention and 48 hours after the intervention
  laboratory test
The level of cholesterol | before the intervention and 48 hours after the intervention
  laboratory test
The level of alanine aminotransferase (ALT) | before the intervention and 48 hours after the intervention
  laboratory test
The level aspartate aminotransferase (AST) | Before the intervention and 48 hours after the intervention
  laboratory test
The level of alkaline phosphatase (ALP) | Before the intervention and 48 hours after the intervention
  laboratory test

SECONDARY OUTCOMES:
The level of anxiety | Before the intervention and after the intervention
  With the history of taking and filling the DASS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tarbiat Modares university, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided